CLINICAL TRIAL: NCT03319641
Title: 68Ga-PSMA-PET/CT Imaging for Locally Advanced, Recurrent and Metastatic Adenoid Cystic Carcinoma or Salivary Duct Carcinoma
Brief Title: PSMA-PET Imaging for Advanced ACC/SDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Adenoid Cystic Carcinoma Research Foundation (Other)
Responsible Party: Principal Investigator, Carla van Herpen, MD, PhD, Radboud University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 104902
Record Dates: First submitted 2017-09-29; First posted 2017-10-24 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Salivary Gland Cancer; Adenoid Cystic Carcinoma; Salivary Duct Carcinoma
Keywords: 68Ga-PSMA; Positron-Emission Tomography; Immunohistochemistry
MeSH Terms: conditions — Salivary Gland Neoplasms; Carcinoma, Adenoid Cystic

STUDY DESIGN:
Intervention Model Description: diagnostic study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSMA-PET/CT scan (Experimental): PSMA-PET/CT imaging in advanced ACC/SDC
  Interventions: Diagnostic Test: PSMA-PET/CT scan

INTERVENTIONS:
Diagnostic Test: PSMA-PET/CT scan — perform a PSMA-PET/CT scan in patients with locally advanced, recurrent and/or metastastic ACC or SDC

SUMMARY:
Diagnostic study which evaluates the level of PSMA expression in patients with locally advanced, recurrent and/or metastatic ACC/SDC of ≥18 years old with 68Ga-PSMA-PET/CT imaging in order to establish whether these patients are eligible for 177Lu-PSMA therapy

DETAILED DESCRIPTION:
Rationale: PSMA is a transmembrane protein, which is expressed on prostate cancers cells, ACC and other malignancies. In prostate cancer, distant metastases can be visualized sensitively and non-invasively with 68Ga-PSMA-PET/CT scans and if the uptake of 68Ga is high enough, patients can be treated with the β-emitting radionuclide 177Lu-PSMA. In the current study, we will evaluate the uptake of 68Ga-PSMA by performing 68Ga-PSMA-PET/CT scans in advanced ACC and SDC patients. If the uptake is high enough, this will form the rationale for a therapeutic study with 177Lu-PSMA in ACC and SDC.

Objective: The primary objective is to evaluate the uptake of 68Ga-PSMA in locally advanced, recurrent and metastatic ACC/SDC by performing 68Ga-PSMA-PET/CT scans. The secondary objectives are to calculate the SUV tumor-to-background ratio and tumor-to-'healthy salivary gland tissue' ratio. To correlate the SUV to the degree of immunohistochemical PSMA expression of the primary tumor on archival tissue, and to establish whether new metastatic lesions are found by 68GA-PSMA-PET/CT imaging.

Study design: Diagnostic study which evaluates the level of PSMA expression in ACC/SDC patients with 68Ga-PSMA-PET/CT imaging in order to establish whether these patients are eligible for 177Lu-PSMA therapy.

Study population: Patients with locally advanced, recurrent or metastatic ACC/SDC of ≥18 years old.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced, recurrent or metastatic ACC/SDC
* Age ≥ 18 years old
* Ability to provide written informed consent

Exclusion Criteria:

* Contra-indication for PET imaging
* Pregnancy
* Breast feeding
* Severe claustrophobia
* Impaired renal function: MDRD <30 ml/min/1,73 m2
* Impaired liver function: AST and ALT ≥ 2.5 x ULN (≥5 x ULN for patients with liver metastases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
uptake of 68Ga-PSMA in ACC and SDC | 0 days
  To evaluate the uptake of 68Ga-PSMA in locally advanced, recurrent and metastatic ACC/SDC by performing 68Ga-PSMA-PET/CT scans

SECONDARY OUTCOMES:
SUV of 68Ga-PSMA in ACC/SDC tumors | 0 days
  SUV of 68Ga-PSMA in ACC/SDC tumors
SUV of 68Ga-PSMA in the background | 0 days
  in order to calculate the SUV tumor to background ratio
correlation of SUV and IHC PSMA-staining | 0 days
  Correlate the tumor uptake (SUV) to the degree of immunohistochemical PSMA expression of the primary tumor on archival tissue
new metastases | 0 days
  To establish whether new metastatic lesions are found by 68GA-PSMA-PET/CT imaging

CONTACTS AND LOCATIONS:
Overall Officials: Carla ML van Herpen, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT03319641/Prot_SAP_000.pdf